CLINICAL TRIAL: NCT00513851
Title: A Phase I Dose Escalation Study of Daily Oral OSI-930 in Patients With Advanced Solid Tumors
Brief Title: Phase 1 Study of OSI-930 in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-930-102
Record Dates: First submitted 2007-08-07; First posted 2007-08-09 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Cancer; Non-small cell lung cancer; Small cell lung cancer; Uterine cancer; Ovarian cancer; Renal cancer; Head and neck cancer; Cervical cancer; Metastatic cancer; Colorectal cancer; Gastrointestinal stromal tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Uterine Neoplasms; Ovarian Neoplasms; Kidney Neoplasms; Head and Neck Neoplasms; Uterine Cervical Neoplasms; Neoplasm Metastasis; Colorectal Neoplasms; Gastrointestinal Stromal Tumors | interventions — OSI 930

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Once Daily Dosing
  Interventions: Drug: OSI-930
- 2 (Experimental): Twice Daily Dosing
  Interventions: Drug: OSI-930

INTERVENTIONS:
Drug: OSI-930 — Oral OSI-930 administered once daily at increasing doses until disease progression or unacceptable toxicity
  Arms: 1
Drug: OSI-930 — Oral OSI-930 administered twice daily at increasing doses until disease progression or unacceptable toxicity
  Arms: 2

SUMMARY:
Open label, phase 1, dose escalation

DETAILED DESCRIPTION:
Multicenter, open-label, phase 1, dose escalation study to determine the maximum tolerated dose on both once daily (QD) and twice daily (BID) schedules.

Patients may continue to receive OSI-930 until one of the following occurs: disease progression, adverse event requiring withdrawal, failure to recover from toxicity despite a 14-day dosing interruption, medical or ethical reasons, patient request, or patient death.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically documented malignancy that is now advanced and/or metastatic and refractory to established forms of therapy or for which no effective therapy exists.

Age >/= 18 years, ECOG PS 0-2, life expectancy >/= 12 weeks Prior chemotherapy is permitted provided that a minimum of 3 weeks has elapsed. Prior tyrosine kinase inhibitor therapy is permitted. Patients must have recovered from any treatment-related toxicities (with some exceptions) prior to registration.

Prior hormonal therapy is permitted provided it is discontinued prior to registration (with the exception of prostate cancer patients who have been on hormone therapy for at least 3 months).

Prior radiation therapy is permitted provided that it did not exceed 25% of bone marrow reserve and patients have recovered from the toxic effects. A minimum of 21 days must have elapsed unless the radiotherapy was palliative and nonmyelosuppressive.

ANC >/= 1.5 x 10^9/L, PLT >/= 100 x 10^9/L; bilirubin </= 1.5 x upper limit of normal (ULN), AST and ALT </= 2.5 x ULN; creatinine </= 1.5 ULN Accessible for repeat dosing and follow-up. Patients must practice effective contraceptive measures throughout the study. Provide written informed consent.

Exclusion Criteria:

Symptomatic brain metastases which are not stable, require steroids, are potentially life-threatening or that have required radiation within the last 28 days.

History of allergic reaction attributed to a similar compound as study drug. Significant cardiac disease unless well controlled, poorly controlled hypertension.

Active or uncontrolled infections of serious illnesses or medical conditions that could interfere with participation.

History of any psychiatric condition that might impair the patient's ability to provide informed consent or participate.

Concurrent anticancer therapy. Use of CYP3A4 inducers/inhibitors during the 14 days prior to first dose. Pregnant or breast-feeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) for both the once daily (QD) and twice daily (BID) dosing schedules and establish a recommended phase 2 dose of OSI-930 | 2.5 years

SECONDARY OUTCOMES:
Safety, Pharmacokinetic profile, Pharmacodynamic relationships, Preliminary antitumor activity | 2.5 years

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Dana-Farber Cancer Institute, Boston, Massachusetts
- Cancer Research UK Professor of Medical Oncology, Sutton, Surrey, United Kingdom